CLINICAL TRIAL: NCT07058779
Title: A Randomized, Double-blind, Placebo-controlled Phase I Clinical Study to Evaluate the Safety, Tolerability, Pharmacokinetic and Pharmacodynamic Characteristics of SSS55 Injection in Healthy Subjects in China
Brief Title: Safety, Tolerability, PK and PD of SSS55 in Healthy Subjects
Status: Not yet recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: Shenyang Sunshine Pharmaceutical Co., LTD. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Sequential | Masking: Quadruple | Purpose: Other
Other Study IDs: SSS55-101
Record Dates: First submitted 2025-05-26; First posted 2025-07-10 (Actual); Last update posted 2025-07-10 (Actual); Status verified 2025-06

CONDITIONS: Safety Issues

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- Low-dose group (Experimental): dose1
  Interventions: Drug: SSS55
- middle-dose group (Experimental): dose 2
  Interventions: Drug: SSS55
- high-dose group (Experimental): dose 3
  Interventions: Drug: SSS55
- Higher-dose group (Experimental): dose 4
  Interventions: Drug: SSS55

INTERVENTIONS:
Drug: SSS55 — SSS55 is an injection targeting complement C3b
  Other Names: SSS55 injection

SUMMARY:
This study was a single-dose, randomized, double-blind, placebo-controlled study of SSS55 injection to evaluate the safety, tolerability, PK characteristics, immunogenicity and preliminary efficacy characteristics of single-dose SSS55 injection in healthy individuals.

DETAILED DESCRIPTION:
This study was a single-dose, randomized, double-blind, placebo-controlled study of SSS55 injection to evaluate the safety, tolerability, PK characteristics, immunogenicity and preliminary efficacy characteristics of single-dose SSS55 injection in healthy individuals.In this trial, four dose groups were preset. The initial dose and dose level were relatively low. Two subjects were planned to be enrolled and only received SSS55 administration. In the subsequent dose group, sentries were set up in each group. In each group, the first two subjects were randomly administered with sentries at a ratio of 1:1 between the test drug SSS55 and the placebo. The sentries were involved in blinding. After the sentries completed the safety assessment 8 days after administration, the remaining subjects in the group were administered in a random ratio between the test drug group and the placebo group.

ELIGIBILITY:
Inclusion Criteria:

1. Healthy subjects aged 18 to 45 years old (including the boundary value), regardless of gender;
2. The subjects voluntarily participated in the clinical trial and signed the informed consent form;
3. Men with a weight of ≥50 kg, women with a weight of ≥45 kg, and those with a body mass index (BMI) ranging from 19 to 28 kg/m2 (including the critical value);
4. Those who underwent vital sign assessment, physical examination, blood routine, urine routine, blood biochemistry, coagulation function, pregnancy examination (for women of childbearing age), 12-lead ECG, chest X-ray/lung CT during screening, and the results showed no abnormalities or the abnormalities had no clinical significance;
5. Be willing to receive the MV-ACYW meningococcal vaccine and pneumococcal vaccine 14 days or more before randomization.

Exclusion Criteria:

* 1) Those with a clear history of drug or food allergies, or a known history of hypersensitivity reactions that are clinically significant to the research intervention measures or related compounds or commonly used antibacterial agents;

  2) Those with a history of any serious clinical diseases in the past or present, including but not limited to those in the digestive system, cardiovascular system, respiratory system, urinary system, musculoskeletal system, endocrine system, immune system, neuropsychiatric system, hematological system, etc. (except those deemed eligible for enrollment by the researcher);

  3) First-degree relatives with a known history of meningococcal infection or a history of meningococcal infection;

  4) Those with contraindications to meningococcal vaccination (with a history of epilepsy or other brain diseases, etc.);

  5) There was or suspected active viral, bacterial, fungal or parasitic infection within 14 days prior to screening, including herpes, shingles or cold sores;

  6) A history of recurrent infections of unknown cause; Or systemic antibiotics (intravenous antibiotics, oral antibiotics, etc., excluding topical application antibiotics) have been used within 90 days before administration;

  7) There is a history of Gilbert syndrome or the researcher assesses that it meets the diagnostic criteria for the disease;

  8) Received treatment with blood products within 6 months prior to administration;

  9) Those who have undergone major surgical operations within 4 weeks prior to administration or have not fully recovered from any previous invasive procedures;

  10) Suffering from syphilis (Treponema pallidum antibody positive) or AIDS (HIV antibody positive), or active hepatitis C (hepatitis C virus antibody positive), or active hepatitis B (hepatitis B surface antigen positive);

  11) A history of malignant tumors in the past or present;

  12) Any drugs (including prescription drugs, over-the-counter drugs, Chinese herbal medicines, etc.) or health supplements have been used within 2 weeks before administration (if determined by the investigator, the time interval from the start of administration of the drug in this trial > Five half-lives, and the corresponding subjects can also be enrolled.

Ages: 18 Years to 45 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 26 (Estimated)
Dates: Start 2025-07 (Estimated); Primary Completion 2026-12 (Estimated); Study Completion 2027-12 (Estimated)

PRIMARY OUTCOMES:
To evaluate the safety and tolerability of a single intravenous infusion of SSS55 injection in healthy adult subjects in China | 22days
  Number of participants with treatment-related adverse events as assessed by CTCAE v4.0

SECONDARY OUTCOMES:
To evaluate the pharmacokinetic (PK) characteristics of SSS55 injection after a single intravenous infusion in healthy adult subjects in China | 22days
  To evaluate the AUC of SSS55 injection
To evaluate the pharmacodynamic characteristics of SSS55 injection after a single intravenous infusion in healthy adult subjects in China | 22 days
  To evaluate the complement3 of SSS55 injection
To evaluate the ADA of SSS55 injection after a single intravenous infusion in healthy adult subjects in China | 22days
  To evaluate the ADA of SSS55 injection

IPD SHARING:
Plan to Share IPD: No